CLINICAL TRIAL: NCT02166892
Title: The Effect of Specially Designed Eating Plates on Self-served Portions and Caloric Intake in Normal Weight and Overweight Children
Brief Title: Specially Designed Eating Plates Effects on Food Intake in Normal Weight and Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dan Nemet, MD (Other)
Responsible Party: Sponsor-Investigator, Dan Nemet, MD, Prof. Dan Nemet. MD, Meir Medical Center
Organization: Meir Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MeirMc0042-14CTIL
Record Dates: First submitted 2014-06-09; First posted 2014-06-18 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: Childhood obesity; Plate; Food consumption
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal weight (Active Comparator): Normal weight children will be served food in two different occasions using two sets of plates (same size). One set will be plane and the second is a specially designed plate that demonstrate the recommended food consumption and portion.
  Interventions: Other: Specially designed plates
- Overweight children (Active Comparator): Overweight children will be served food in two different occasions using two sets of plates (same size). One set will be plane and the second is a specially designed plate that demonstrate the recommended food consumption and portion.
  Interventions: Other: Specially designed plates

INTERVENTIONS:
Other: Specially designed plates

SUMMARY:
Previous studies demonstrated that children served themselves more food when using larger plates and bowels. The purpose of this study is to evaluate if self-served portions and caloric intake in normal weight and overweight children will be influenced by a specially designed eating plates compared to similar size normal plates.

DETAILED DESCRIPTION:
40 normal weight and 40 overweight kindergarden and elementary school children will participate in this study.

Anthropometric measurements: weight, height, BMI and BMI percentiles will be measured and calculated for each participant.

The participants will take part in two non-exercise activities at the 'sport and health center for children and adolescence'. At the end of each activity, a lunch buffet that contains all food ingredients will be served. During one meeting the children will be handed a regular plate and at the second meeting they will be handed a specially designed plate (with marking of the recommended meal composition and portion).

The amount and composition of food on the plates will be assessed by weighing and photography before and after eating and analysed to report macronutrient consumption by a dietitian. The meetings for normal weight children will be separated from the overweight children.

ELIGIBILITY:
Inclusion Criteria:

* Over weight / obese children
* Normal weight children

Exclusion Criteria:

* Organic disease that cause obesity
* Underweight children (BMI percentiles < 5)

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Caloric intake | Up to 1 hour after food serving
  The amount of food and drink consumed by the children will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel